CLINICAL TRIAL: NCT03747965
Title: Phase I Study of CRISPR-Cas9 Mediated PD-1 Gene-knocked Out Mesothelin-directed CAR-T Cells With the Conditioning Regimen of Paclitaxel and Cyclophosphamide in Mesothelin Positive Multiple Solid Tumors
Brief Title: Study of PD-1 Gene-knocked Out Mesothelin-directed CAR-T Cells With the Conditioning of PC in Mesothelin Positive Multiple Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, Director, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2017-074-01
Record Dates: First submitted 2018-11-19; First posted 2018-11-20 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Solid Tumor, Adult

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mesothelin-directed CAR-T cells infusion (Experimental): Patients receive mesothelin-directed CAR-T cells infusion with dose escalation will occur using a standard "3+3" dose escalation approach, beginning in dose level I with dose cohorts and rules for escalation and de-escalation.
  Interventions: Biological: Mesothelin-directed CAR-T cells

INTERVENTIONS:
Biological: Mesothelin-directed CAR-T cells — Cells will be infused one day after the completion of conditioning regimen of paclitaxel and cyclophosphamide

SUMMARY:
Multiple solid tumors have positive targets of mesothelin expressed on the surfaces of the tumor cells, the investigators use the technique of CRISPR-Cas9 to knocked out the PD-1 of the chimeric antigen receptor (CAR) T cells with the combination of Pretreatment by Paclitaxel and Cyclophosphamideto to effect the immuno-microenvironment around tumors.

DETAILED DESCRIPTION:
1. To evaluate the feasibility and safety of CRISPR-Cas9 mediated PD-1 gene-knocked out chimeric antigen receptor (CAR) T cells in patients with mesothelin positive multiple solid tumors.
2. To evaluate the duration and in vivo persistence of transferred CAR-T cells.
3. To observe and measure anti-tumor responses for patients with detectable mesothelin positive tumor lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed with mesothelin positive multiple solid tumors, especially in Pancreatic cancer, cholangiocarcinoma cancer and ovarian cancer .
2. Failure of at least one prior standard of care chemotherapy for advanced stage disease.
3. Subjects must have measureable disease as defined by RECIST 1.1 criteria or modified RECIST criteria.
4. Patients > 18 years of age.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Life expectancy > 12 weeks.
7. Satisfactory organ and bone marrow function as defined by the following (of note, the minimal blood counts should be in the absence of transfusion or cytokine support):

   i.Absolute neutrophil count > 1,000/μl ii.Platelets >75,000/μl iii.Hemoglobin > 9 g/dL iv.Bilirubin < 2 times of the institutional normal upper limit unless secondary to bile duct obstruction by tumor v.Creatinine < 1.5 times of the institutional normal upper limit vi.Albumin ≥2 vii.Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) < 5 times of the institutional normal upper limit viii.Cardiac ejection fraction of >45% as measured by resting echocardiogram, with no significant pericardial effusion ix.Normal lung function
8. Blood coagulation parameters: PT such that international normalized ratio (INR) is ≤ 1.5 and a PTT < 1.2 times of the upper limit of normal unless the patient is therapeutically anti-coagulated for history of cancer-related thrombosis and has stable coagulation parameters.
9. Ability to understand and the willingness to provide written informed consent.
10. Male and Female subjects of reproductive potential agree to use approved contraceptive methods (e.g. birth control pills, barrier device, intrauterine device, abstinence) and abstain from other methods of conception during the study and for 6 months following the study cell infusion or proof of sterility.

Exclusion Criteria:

1. Patients with moderate or higher hydrothorax and abdominal effusion, which are difficult to control by conventional treatment and require continuous catheter drainage;
2. Either of the following virological tests is positive: HIV;HCV.HBsAg;Positive HBV DNA copy number was detected simultaneously (quantitative detection was 5 x 10^2 copies/ml).RPR or TPPA positive;
3. Other malignant tumors, with the exception of basal cell carcinoma of the skin, superficial cervical cancer, bladder cancer, and prostate cancer(PSA value < 1.0) that do not require further treatment;
4. Accompanied by central metastasis;
5. Severe, uncontrollable comorbidities that may affect program compliance or interpretation of interference results, or any serious medical conditions that may affect the safety of the subject (such as uncontrollable heart disease, hypertension, active virus, bacterial infection or uncontrollable systemic fungal infection);
6. Active autoimmune diseases (including but not limited to systemic lupus erythematosus, sjogren's syndrome, rheumatoid arthritis, psoriasis, multiple sclerosis, inflammatory bowel disease, etc.) need to be treated with immunosuppressive therapy within 4 weeks before enrollment, with the exception of thyroid hormone replacement therapy;
7. Subjects are receiving immunosuppressive, glucocorticoid (systemic or local) therapy (dose >10mg/ day prednisone or other equivalent hormones), and continue to use it within 2 weeks before enrollment;
8. With the history of organ transplantation;
9. Subjects who were given the last treatment less than 4 weeks before the initial treatment or participated in other relevant clinical study subjects at the same time;
10. With the history of gene therapy;
11. During the period of first study, live vaccines were administered within 4 weeks before PBMC collection;
12. People who have a history of psychotropic drug abuse and are unable to get rid of it or have a history of mental disorders;
13. Life-threatening allergic, hypersensitive, or intolerant reactions to GC008t preparations or their excipients (including DMSO) are known;
14. Hemorrhagic and thrombotic tendencies:3 months prior to study drug treatment for the first time there have been significant clinical significance of bleeding symptoms or have a definite bleeding tendency, such as gastrointestinal bleeding, bleeding ulcers, coagulant function abnormality (PT > 16 s, APTT, TT > > 43 s 21 s, FIB < 2 g/L), there is tendency of inherited or acquired bleeding and thrombosis (such as hemophilia, blood coagulation dysfunction, thrombocytopenia, the splenic function, etc.), were treated with thrombolysis and anticoagulation, 6 months prior to study drug treatment for the first time move/enous thromboembolism events,Such as cerebral vascular diseases (including cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism;
15. Other severe, acute or chronic medical or mental illnesses that may increase the risk of participating in the study or may interfere with the interpretation of the results, according to the researchers.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Study of related adverse events | 24 weeks
  Grade 3 or severer signs/symptoms, toxicities and clinical

SECONDARY OUTCOMES:
Clinical responses of mesothelin-directed CAR T cells infusion | 24 weeks
  Disease control rate(DCR)

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Han, Dr, Study Director — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No